CLINICAL TRIAL: NCT04434469
Title: An Open-Label, Multicenter, Phase I Trial Evaluating The Safety And Pharmacokinetics Of Escalating Doses Of RO7297089 In Patients With Relapsed Or Refractory Multiple Myeloma
Brief Title: A Study Evaluating The Safety And Pharmacokinetics Of Escalating Doses Of RO7297089 In Patients With Relapsed Or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO41582
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Refractory Multiple Myeloma; Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm A Flat Dose Escalation: RO7297089 (Experimental): Participants in Arm A will receive the target dose of RO7297089 as a flat dose at each scheduled study drug administration visit
  Interventions: Drug: RO7297089
- Arm B Split Dose Escalation: RO7297089 (Experimental): Participants in Arm B will receive the first target dose of RO7297089 as a split dose divided over two days (Days 1 and 2). The full target dose will be administered at subsequent study drug administration visits.
  Interventions: Drug: RO7297089
- Arm C Step Dose Escalation: RO7297089 (Experimental): No participants enrolled. Enrollment for the GO41582 study was stopped in July 2021 due to limited activity as a single agent which did not meet the Sponsor's internal criteria for further clinical development.
  Interventions: Drug: RO7297089
- Phase I Expansion Stage: RO7297089 (Experimental): No participants enrolled. Enrollment for the GO41582 study was stopped in July 2021 due to limited activity as a single agent which did not meet the Sponsor's internal criteria for further clinical development.
  Interventions: Drug: RO7297089

INTERVENTIONS:
Drug: RO7297089 — RO7297089 will be given via intravenous (IV) infusion

SUMMARY:
This is a first-in-human Phase I, open-label, multicenter, global, dose-escalation study designed to evaluate the safety, tolerability, and pharmacokinetics of RO7297089 and make a preliminary assessment of anti-tumor activity in patients with R/R MM for whom no established therapy for MM is appropriate and available or who are intolerant to those established therapies.

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* R/R MM for which no established therapy for MM is appropriate and available or be intolerant to those established therapies
* Measurable disease

Exclusion criteria:

* Prior use of any monoclonal antibody, radioimmunoconjugate, or antibody-drug conjugate for the treatment of cancer within 4 weeks before first RO7297089 infusion
* Prior treatment with systemic immunotherapeutic agents within 12 weeks or 5 half-lives of the drug, whichever is shorter, before first RO7297089 infusion
* Prior treatment with CAR-T therapy within 90 days before first study drug administration
* Treatment with any chemotherapeutic agent, or treatment with any other anti-cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first RO7297089 infusion
* Autologous stem cell transplantation within 100 days prior to first RO7297089 infusion
* Allogeneic stem cell transplantation within 180 days prior to first RO7297089 infusion or requiring immunosuppression for treatment or prophylaxis of graft versus host disease
* Primary or secondary plasma cell leukemia
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection requiring treatment with IV anti-microbial therapy within 14 days prior to first RO7297089 infusion
* Significant cardiovascular disease
* Current CNS involvement by MM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Australia (5):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - LIVERPOOL HOSPITAL; HAEMATOLOGY; Ingham Institute for Medical Research, Liverpool, New South Wales
  - Royal Adelaide Hospital; Haematology Clinical Trials, Adelaide, South Australia
  - St. Vincent's Hospital Melbourne, Fitzroy, South Australia
  - Peter Mac Callum Cancer Center, East Melbourne, Victoria
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Denmark (2):
  - Rigshospitalet, København Ø
  - Vejle Sygehus; Onkologisk Afdeling, Vejle
- Oslo Universitetssykehus HF; Ullevål sykehus, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

REFERENCES:
- [Derived] Plesner T, Harrison SJ, Quach H, Lee C, Bryant A, Vangsted A, Estell J, Delforge M, Offner F, Twomey P, Choeurng V, Li J, Hendricks R, Ruppert SM, Sumiyoshi T, Miller K, Cho E, Schjesvold F. Phase I Study of Safety and Pharmacokinetics of RO7297089, an Anti-BCMA/CD16a Bispecific Antibody, in Patients with Relapsed, Refractory Multiple Myeloma. Clin Hematol Int. 2023 Mar;5(1):43-51. doi: 10.1007/s44228-022-00023-5. Epub 2023 Jan 19. PMID 36656461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a screening period of up to 28 days and a minimum follow-up period of 90 days after treatment. Following confirmation of eligibility, patients received RO7297089 by intravenous (IV) infusion. Patients were enrolled in two stages: a dose escalation stage and an expansion stage.
Groups:
- Dose Escalation Cohort 1: RO7297089: Participants in Arm A received 60 mg dose of RO7297089 as a flat dose at each scheduled study drug administration visit
- Dose Escalation Cohort 2: RO7297089: Participants in Arm A received 180 mg dose of RO7297089 as a flat dose at each scheduled study drug administration visit
- Dose Escalation Cohort 3: RO7297089: Participants in Arm A received 360 mg dose of RO7297089 as a flat dose at each scheduled study drug administration visit
- Dose Escalation Cohort 4: RO7297089: Participants in Arm A received 1080 mg dose of RO7297089 as a flat dose at each scheduled study drug administration visit
- Dose Escalation Backfill Cohort 4: RO7297089: Participants in Arm B received the 1080 mg dose of RO7297089 as a split dose divided over two days (Days 1 and 2). The full target dose wasadministered at subsequent study drug administration visits.
- Dose Escalation Cohort 5: RO7297089: Participants in Arm B received the 1850 mg dose of RO7297089 as a split dose divided over two days (Days 1 and 2). The full target dose was administered at subsequent study drug administration visits.
Period: Overall Study
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Started | 3 | 5 | 4 | 6 | 6 | 3
Completed (Alive: In Follow-up) | 0 | 1 | 0 | 1 | 0 | 0
Not Completed | 3 | 4 | 4 | 5 | 6 | 3
Not completed — Death | 2 | 3 | 2 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Study terminated by sponsor | 1 | 1 | 1 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089 | Total
Number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 3 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 4 | 3 | 5 | 2 | 17
  >=65 years | 3 | 2 | 0 | 3 | 1 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (1.2) | 62.6 (9.2) | 54.3 (9.4) | 63.0 (4.1) | 60.2 (6.3) | 65.7 (7.4) | 61.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 3 | 2 | 0 | 8
  Male | 3 | 4 | 2 | 3 | 4 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 3 | 5 | 3 | 3 | 22
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 3 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 3 | 5 | 6 | 3 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Including Dose Limiting Toxicities (DLTs)
Description: Adverse event severity graded according to NCI CTCAE v5.0
Time Frame: Baseline up to 1 year 7 months
Population: Safety-Evaluable Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 3
Percentage of Participants | 100 | 100 | 75 | 100 | 83.3 | 100

2. Secondary Outcome: Time to Maximum Concentration Observed (Tmax) of RO7297089
Time Frame: Cycle 1 Day 1
Population: Cohorts reported with participants excluded from descriptive statistics due to not receiving the full dose:
  Cohort 2: 1 participant Cohort 3: 1 participant Cohort 4A: 2 participants Cohort 4B reported with 1 participant excluded from descriptive statistics due to apparent outlier and 1 participant due to or missing sample.
Measure: Median (Full Range); unit: EOI, day
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 4 | 3
EOI, day | 0.25 [0.08 to 0.25] | 0.17 [0.08 to 0.25] | 0.08 [0.08 to 0.08] | 0.25 [0.25 to 0.25] | 1.08 [1.08 to 1.17] | 1.08 [1.08 to 2.11]

3. Secondary Outcome: Area Under the Curve (AUC) of RO7297089
Time Frame: Cycle 1 Day 1
Population: Only those participants who received full dose were included in the results summary
Measure: Geometric Mean (Standard Deviation); unit: ug/mL*day
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 4 | 3
ug/mL*day | 12.7 (26.3) | 78.7 (31.3) | 280 (73.6) | 1347 (NA) — Only 1 participant analyzed | 1046 (28.0) | 1920 (25.4)

4. Secondary Outcome: Maximum Concentration Observed (Cmax) of RO7297089
Time Frame: Cycle 1 Day 1, Cycle 2 Day 8
Population: Only those participants who received full dose were included in the results summary
Measure: Geometric Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 4 | 3
ug/mL
  C1D1 | 7.79 (21.6) | 40.9 (46.3) | 95.9 (35.8) | 314 (NA) — Only 1 participant analyzed | 305 (15.5) | 404 (12.4)
  C2D8 | 9.50 (24.1) | 48.6 (23.6) | 153 (47.5) | 394 (NA) — Only 1 participant analyzed | 541 (38.9) | 966 (24.7)

5. Secondary Outcome: Minimum Concentration Observed (Cmin) of RO7297089
Time Frame: Cycle 1 Day 1, Cycle 2 Day 8
Population: Only those participants who received full dose were included in the results summary
Measure: Geometric Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 4 | 3
ug/mL
  C1D1 | 0.19 (22.3) | 0.96 (42.5) | 9.19 (500) | 140 (NA) — Only 1 participant analyzed | 81.3 (85.1) | 197 (32.6)
  C2D8: number analyzed (Participants) | 3 | 1 | 3 | 1 | 4 | 3
  C2D8 | 0.25 (39.9) | 2.99 (NA) — Only 1 participant analyzed | 19.7 (372) | 163 (NA) — Only 1 participant analyzed | 207 (90.0) | 450 (40.2)

6. Secondary Outcome: Half-life (t1/2) of RO7297089
Time Frame: Cycle 1 Day 1
Population: Only those participants who received full dose were included in the results summary
Measure: Geometric Mean (Standard Deviation); unit: day
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 4 | 3
day | 1.39 (8.33) | 1.25 (14.9) | 2.39 (89.5) | 6.73 (NA) — Only 1 participant analyzed | 4.22 (83.7) | 6.52 (24.5)

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as a Stringent Complete Response (Scr), Complete Response (CR), Very Good Partial Response (VGPR) or Partial Response (PR) as determined by the Investigator according to International Myeloma Working Group (IMWG) Uniform Response Criteria
Time Frame: Baseline up to approximately 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 3
Participants
  Partial Response | 0 | 0 | 0 | 1 | 0 | 1
  Minimal Response | 0 | 0 | 1 | 0 | 1 | 0
  Stable disease | 1 | 2 | 3 | 4 | 4 | 2
  Progressive disease | 2 | 2 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 1 year and 7 months
Arm/Group | Dose Escalation Cohort 1: RO7297089 | Dose Escalation Cohort 2: RO7297089 | Dose Escalation Cohort 3: RO7297089 | Dose Escalation Cohort 4: RO7297089 | Dose Escalation Backfill Cohort 4: RO7297089 | Dose Escalation Cohort 5: RO7297089
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/5 | 2/4 | 2/6 | 2/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/5 | 3/4 | 5/6 | 4/6 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 5/5 | 3/4 | 6/6 | 5/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Cohort 1: RO7297089 (N=3) | Dose Escalation Cohort 2: RO7297089 (N=5) | Dose Escalation Cohort 3: RO7297089 (N=4) | Dose Escalation Cohort 4: RO7297089 (N=6) | Dose Escalation Backfill Cohort 4: RO7297089 (N=6) | Dose Escalation Cohort 5: RO7297089 (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Cohort 1: RO7297089 (N=3) | Dose Escalation Cohort 2: RO7297089 (N=5) | Dose Escalation Cohort 3: RO7297089 (N=4) | Dose Escalation Cohort 4: RO7297089 (N=6) | Dose Escalation Backfill Cohort 4: RO7297089 (N=6) | Dose Escalation Cohort 5: RO7297089 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 3 (5) | 3 (4) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calcium ionised increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04434469/Prot_SAP_000.pdf